CLINICAL TRIAL: NCT01065376
Title: The Influence of Dopamine Agonist Cabergoline on Oocyte Maturation in Women Undergoing Assisted Reproduction
Brief Title: The Influence of Dopamine Agonist Cabergoline on Oocyte Maturation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Jiann-Loung Hwang, Shin-Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKH-8302-99-DR-28
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-04

CONDITIONS: In Vitro Fertilization
Keywords: IVF; OHSS; cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- on the day of hCG (Experimental): cabergoline administration for 8 days on the day of hCG.
  Interventions: Procedure: the timing cabergoline administration
- on the day after oocyte retrieval (Experimental): cabergoline administration for 8 days on the day after oocyte retrieval
  Interventions: Procedure: the timing cabergoline administration

INTERVENTIONS:
Procedure: the timing cabergoline administration — received 0.5 mg oral cabergoline per day for 8 days on the day of hCG
  Arms: on the day of hCG
Procedure: the timing cabergoline administration — received 0.5 mg oral cabergoline per day for 8 days on the day after oocyte retrieval
  Arms: on the day after oocyte retrieval

SUMMARY:
The dopamine agonist cabergoline inhibits phosphorylation of the vascular endothelial growth factor receptor-2(VEGFR-2), which prevent vascular endothelial growth factor (VEGF) overexpression and reduce the severity of Ovarian hyperstimulation syndrome. However, VEGF plays an important role in the growth and maintenance of ovarian follicle and developing embryo by mediating angiogenesis.This study was designed to analyze whether the timing cabergoline administration on the day of human chorionic gonadotropin (hCG) injection or after oocytes retrieved affects the oocyte maturation and outcome of assisted reproduction treatment.

DETAILED DESCRIPTION:
BACKGROUND:Ovarian hyperstimulation syndrome (OHSS) is the most serious complication of ovulation induction. It results from increased vascular permeability caused by ovarian hypersecretion of VEGF), which activates its receptor-2. The dopamine agonist cabergoline inhibits phosphorylation of the receptor VEGFR-2, which prevent VEGF overexpression and reduce the severity of OHSS. However, VEGF plays an important role in the growth and maintenance of ovarian follicle and developing embryo by mediating angiogenesis. In human, cabergoline averts OHSS, but a possible detrimental effect on oocyte maturation has not been explored. This study was designed to analyze whether the timing cabergoline administration on the day of hCG injection or after oocytes retrieved affects the oocyte maturation and outcome of assisted reproduction treatment.

PURPOSE: To assess whether the timing cabergoline administration affects metaphase II oocytes numbers, embryo quality, pregnancy outcome and the incidence of OHSS.

METHODS: A prospective randomized study was designed to evaluate the possible of cabergoline affect on oocyte maturation. Women (n=120) under controlled ovarian hyperstimulation with the risk of OHSS (Estradiol(E2)>4000 pg/ml, or >18 follicle, >11 mm development) randomized into two groups. Group I (n=60) received 0.5 mg oral cabergoline per day for 8 days on the day of hCG. Group II (n=60) received 0.5 mg oral cabergoline per day for 8 days on the day after oocyte retrieval immediately.

ANTICIPATED RESULTS: No significant differences were seen in the number of metaphase II oocytes, the embryo quality, the pregnancy rate and the incidence of OHSS.

ELIGIBILITY:
Inclusion Criteria:

* the risk of ovarian hyperstimulation syndrome development

Exclusion Criteria:

* allergic to cabergoline

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
number of metaphase II oocytes | one year

SECONDARY OUTCOMES:
embryo quality | one year
pregnancy rate | one year
The incidence of OHSS | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jiann-Loung Hwang, MD, Study Chair — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Shin-Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan